CLINICAL TRIAL: NCT05355220
Title: Effects of Silver Spike Point Therapy on Pelvic Girdle Pain and Functional Activities in Pregnancy
Brief Title: Effects of Silver Spike Point Therapy on Pelvic Girdle Pain PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0506 Maida
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Pelvic Girdle Pain
Keywords: Pelvic girdle pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- silver spike point Therapy Group (Experimental): One group will receive electrotherapy (silver spike point) for 10 mints along with conservative managment
  Interventions: Device: Silver Spike Point Therapy (SSPT)
- Conservative treatment group (Active Comparator): 2nd group will receive strengthening, stretching and stabilization exercises for prlvic girlde
  Interventions: Other: Conservative Managment

INTERVENTIONS:
Device: Silver Spike Point Therapy (SSPT) — Silver Spike Point Therapy (SSPT) means passing an electric current through the skin surface with the triangle spike silver coated metal electrode. SSPT was reported by Hyoto and Kitade in Edinburg, Scotland. 3rd World Congress on Pain in 1981; It has a number of advantages over traditional narcotic medication in pelvic girdle pain management. It does not depress the cardiovascular, respiratory, or the metabolic systems and has no apparent effect on the sensorium
  Arms: silver spike point Therapy Group
Other: Conservative Managment — 2 sets of 10 repetitions Bridging, Cat & cow exercises, Back press exercises, stretching of hip external rotators and extensors 20 sec / stretch
  Arms: Conservative treatment group

SUMMARY:
The aim of this study is to determine the effects of Silver Spike Point Therapy (SSPT) therapy on pelvic girdle pain and functional activities in pregnancy.The finding of this study will help to establish the role of SSPT therapy to relieve pelvic girdle pain in pregnant females along with exercises. SSP for pelvic girdle pain management can prove to be a useful method. The findings of this study can play a role to establish more rigorous treatment plans for pelvic girdle pain in the pregnant population in the future.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial that will investigate the effectiveness of silver spike point therapy and manual therapy in subjects with pregnancy-related pelvic girdle pain. Subjects with pregnancy-related pelvic girdle pain meeting the predetermined inclusion & exclusion criteria will be divided into two groups using the lottery method. Pre-assessment will be done using NPRS and PGPQ as subjective measurements and PSFS as objective measurements. Subjects in one group will be treated with silver spike point therapy and manual therapy, the other will be treated with manual therapy only. Each subject will receive 10 treatment sessions, with 05 treatment sessions per week. Post-treatment reading for NPRS, PGPQ, and PSFS will be recorded after the end of the 10th treatment session. Recorded values will be analyzed for any significant difference between pre and post-treatment values SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 20 to 40 years of age
* Healthy pregnancy
* 14 to 38 weeks gestation
* Expecting a singleton fetus
* 2 out of 3 tests positive for PGP according to European guidelines for
* pelvic girdle pain"(Posterior pelvic pain provocation (P4), Patrick's Faber, Modified Trendelenburg's test)

Exclusion Criteria:

* High-risk pregnancy, Caudaequina Syndrome, Trauma, or spinal surgical history.
* Inflammatory, infective, metabolic, neoplastic, or degenerative conditions.
* Sensory symptoms associated with disc herniation or compressive spinal lesion.
* Any contraindication to exercise.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS): | 2 weeks
  Pain intensity is frequently measured on an 11-point pain intensity numerical rating scale (PI- NRS), where 0=no pain and 10=worst possible pain. However, it is difficult to interpret the clinical importance of changes from baseline on this scale (such as a 1- or 2-point change)
Pelvic Girdle Pain Questionnaire (PGPQ): | 2 weeks
  The Pelvic Girdle Questionnaire (PGQ) is a condition-specific measure for women with pelvic girdle pain (PGP). The PGQ includes items relating to activity/participation and bodily symptoms and has reliability, validity, and feasibility for use in research and clinical practice
Patient specific Functional Scale (PSFS) | 2 weeks
  Patient Specific Functional Scale was developed by Stratford et al 1995 as a self-report outcome measure of function that could be used in patients with varying levels of independence. The aim of PSFS is to provide clinicians with a valid, reliable, responsive andefficient outcome measure that would be easy
  to use and applicable to a large number of clinical presentations. Patient- Specific Functional Scale is an efficient and valid measure for assessing
  disability and change in disability in persons with musculoskeletal diseases

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Hamza Hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdul Salam K. A Comparative study to Assess the Effectiveness of Combined Tens andExercises over Exercise Alone for Sacroiliac Joint Pain in Pregnancy: College of Physiotherapy,Trinity Mission and Medical Foundation, Madurai; 2011.
- [Background] Casagrande D, Gugala Z, Clark SM, Lindsey RW. Low Back Pain and Pelvic Girdle Pain in Pregnancy. J Am Acad Orthop Surg. 2015 Sep;23(9):539-49. doi: 10.5435/JAAOS-D-14-00248. Epub 2015 Aug 13. PMID 26271756
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Background] Elden H, Ostgaard HC, Fagevik-Olsen M, Ladfors L, Hagberg H. Treatments of pelvic girdle pain in pregnant women: adverse effects of standard treatment, acupuncture and stabilising exercises on the pregnancy, mother, delivery and the fetus/neonate. BMC Complement Altern Med. 2008 Jun 26;8:34. doi: 10.1186/1472-6882-8-34. PMID 18582370
- [Background] Stuge B, Laerum E, Kirkesola G, Vollestad N. The efficacy of a treatment program focusing on specific stabilizing exercises for pelvic girdle pain after pregnancy: a randomized controlled trial. Spine (Phila Pa 1976). 2004 Feb 15;29(4):351-9. doi: 10.1097/01.brs.0000090827.16926.1d. PMID 15094530
- [Background] Lee KS, Kim YH, Min KH, Yoo HK, Hwang YH, Chung CK, et al. Clinical Study of thePostperative Pain Management with Silver Spike Point Electro-therapy. Korean Journal of Anesthesiology. 1985;18(1):63-70.
- [Background] Sawada T, Tateyama N, Ikeda T, Ishimaru K. The Effect on Muscle Hardness of Acupuncture Stimulation Using Low-reactive Level Laser Therapy and Silver Spike Point Therapy, along with Stretching. Laser Ther. 2020 Jul 17;29(1):41-46. doi: 10.5978/islsm.20-OR-04. PMID 32903997
- [Background] Yi D-H, Kim B-R, Hur Y-J, Kim D-H, Shim S-Y, Yim J-E. Convergence of Acupoint andElectrical Stimulation Therapy for Blood Flow and Pain Threshold. Journal of the Korea Convergence Society. 2019;10(6):79-87.
- [Background] Taguchi R. Acupuncture anesthesia and analgesia for clinical acute pain in Japan. Evid Based Complement Alternat Med. 2008 Jun;5(2):153-8. doi: 10.1093/ecam/nem056. PMID 18604250
- [Background] Xu H, Ryan J, Li K. Clinical Investigation into the effectiveness of needleless acupuncture inthe management of the symptoms of osteoarthritis of the knee: a preliminary, single-blind and sham- controlled study. Australian Journal of Acupuncture and Chinese Medicine. 2007;2(2):9-15.
- [Background] Ishimaru K, Kawakita K, Sakita M. Analgesic effects induced by TENS and electroacupuncture with different types of stimulating electrodes on deep tissues in human subjects. Pain. 1995 Nov;63(2):181-187. doi: 10.1016/0304-3959(95)00030-V. PMID 8628583